CLINICAL TRIAL: NCT04819425
Title: "Comparison of Two Methods of Securing Endotracheal Tubes in Intensive Care : Elastic Adhesive Strips vs Lace In A Protective Sheath. A Randomized Multicenter, Cluster and Crossover Controlled Study. FIXATUB"
Brief Title: "Comparison of Two Methods of Securing Endotracheal Tubes in Intensive Care : Elastic Adhesive Strips vs Lace In A Protective Sheath."
Acronym: FIXATUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD032-20
Record Dates: First submitted 2021-03-19; First posted 2021-03-29 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Intubation Complication
Keywords: Endotracheal Tube; Securement; Facial skin tear; Lip ulcer; Critical care

STUDY DESIGN:
Intervention Model Description: Cluster and Crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic Adhesive Strips (Experimental): Endotracheal tube fixed by elastic adhesive tape (Tensoplast type adhesive tape):
  The adhesive tape will be attached to the patient's face (opposite side to the endotracheal tube) and then two turns around the endotracheal tube will be made. The rest of the adhesive tape will be attached to the other side of the face (side of the endotracheal tube).
  The laminated tape will be kept on the adhesive tape until it passes over the neck in order to avoid adhering to the hair.
  Finally, the end of the adhesive tape will be replaced on the part already attached to the patient.
  It will be changed daily and after stain or examinations if necessary.
  Interventions: Device: Elastic Adhesive Strips
- Lace in A Protective Sheath (Active Comparator): A loop is made with the lace then the endotracheal tube is passed through the loop. The loop is tightened by pulling each side on the remaining cords and a knot is made on one side of the fastener.
  It will be changed daily and after stain or examinations if necessary.
  Interventions: Device: Lace in A Protective Sheath

INTERVENTIONS:
Device: Elastic Adhesive Strips — Securement of Endotracheal tube with Elastic Adhesive Strips
  Arms: Elastic Adhesive Strips
Device: Lace in A Protective Sheath — Securement of Endotracheal tube with Lace in A Protective Sheath
  Arms: Lace in A Protective Sheath

SUMMARY:
Every year, in France, nearly 100,000 patients hospitalized in intensive care more than 48 hours require invasive respiratory assistance via an endotracheal tube.

Appropriate tube fixation is essential to ensure effective ventilation while minimizing potential complications such as accidental extubations. However, the fixation system chosen may lead to peribuccal lesions such as bedsores, shearing or cutaneous-mucous tear. These lesions are painful for patients and often unsightly as scar may remain.

There are no formal recommendations for the use of any type of fixing system. Thus, systems used to secure the endotracheal tube vary from one ICU to another.

The objective of this study is to demonstrate that the fixing strategy by elastic adhesive tape reduces the risk of developing a peribuccal lesion during the time of the endotracheal tube's maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in Intensive Care Unit
* Age over 18
* Intubation for estimated duration > 48h
* Patient treated with vasopressors
* Patient or relative who received the information and are not opposed to study participation or patient included under the emergency procedure in the absence of contactable family members.

Exclusion Criteria:

* Pre-existing face lesions at ICU admission along the path of the endotracheal tube fixing.
* Admitted patient already intubated upon transfer from another ICU
* Nasotracheal intubation
* Patient in isolation for suspected COVID or clinically proven COVID
* Admitted tracheotomized patient
* Pregnant, nursing, parturient woman
* Lack of social security affiliation
* Moribund
* Incapable major (under guardianship, curatorship)
* Patient deprived of liberty by court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Peribuccal lesion | up to 10 days after intubation
  Appearance of at least one peribuccal lesion during the first 10 days of maintaining the endotracheal tube inserted orally.
  Presence of peribuccal lesion will be validated on picture by an independent review committee.
  The picture will be taken daily without the visible fixing system (blind maintained for the adjudication committee) from J0 to J10 at the site of the endotracheal tube.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa ZINZONI, Principal Investigator — CHD Vendée
Locations (13):
- France (13):
  - Centre Hospitalier d'Angoulême, Angoulême
  - CH Victor Dupouy, Argenteuil
  - Centre Hopitalier La Rochelle, La Rochelle
  - Centre Hospitalier Le Mans, Le Mans
  - Groupe Hospitalier Bretagne Sud, Lorient
  - CHU Nantes Hôtel Dieu, Nantes
  - Centre Hospitalier Régional d'Orléans, Orléans
  - CHI Poissy - Saint-Germain-en-Laye, Poissy
  - CHU de Poitiers, Poitiers
  - Hôpital Nord Laennec, Saint-Herblain
  - CH Saint-Nazaire, Saint-Nazaire
  - CHU La Réunion GHSR, Saint-Pierre
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zinzoni V, Planche L, Le Potier S, Robin L, Le Parco C, Terrat P, Leroyer MH, Atger R, Dauvergne JE, Muller L, Fontaine L, Morand C, Dennemont P, Paillard O, Vastral S, Dardaine B, Le Guillou S, Maquigneau N, Martin S, Lacherade JC. Impact of two endotracheal tube fixation on the incidence of peri-oral lesions: Elastic adhesive strips versus cord in a protective sheath. Study protocol for a cluster cross-over randomized trial. PLoS One. 2024 Feb 8;19(2):e0297349. doi: 10.1371/journal.pone.0297349. eCollection 2024. PMID 38330026